CLINICAL TRIAL: NCT01442493
Title: Reengineering Methadone Treatment: A Randomized Clinical Trial
Brief Title: Reengineering Methadone Treatment Study of Patient-centered Methadone Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R01DA015842 (NIH)
Record Dates: First submitted 2011-09-07; First posted 2011-09-28 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Opiate Dependence
Keywords: Methadone Treatment; Opiate dependence; Services research
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-Centered Methadone Treatment (Experimental): Patient-Centered Methadone Treatment alters the rules and staff roles in methadone treatment as usual in an attempt to increase treatment retention and improve patient outcomes.
  Interventions: Other: Patient-Centered Methadone Treatment
- Methadone Treatment as Usual (Active Comparator): Methadone treatment provided as usual in the U.S.
  Interventions: Other: Methadone Treatment as usual

INTERVENTIONS:
Other: Patient-Centered Methadone Treatment — Unlike in treatment as usual, counseling will be encouraged but not required and counselors will be responsible for enforcing the clinic's rules. The rules will be enforced by the Clinical Director. Clinic rules will be modified such that involuntary discharge from treatment will be a rare event.
  Arms: Patient-Centered Methadone Treatment
Other: Methadone Treatment as usual — Counseling will be required and counselors will enforce the usual clinic rules. Involuntary discharge may occur for ongoing drug use or rule infractions as usually occurs in the clinic.
  Arms: Methadone Treatment as Usual

SUMMARY:
The purpose of the study is to determine whether a change in the rules and staff roles in methadone treatment programs will result in greater lengths of stay in treatment and lower rates of heroin and cocaine use, crime and HIV-risk behavior as compared to methadone treatment as usual.

DETAILED DESCRIPTION:
Early drop-out and premature discharge from methadone treatment is common in the United States and may be associated with drug use and its associated problems. The purpose of this study is to evaluate the effectiveness of a novel approach to the organization methadone treatment in which the patient rules and staff roles of the clinic will be modified for study participants as compared to patients receiving standard methadone treatment.

ELIGIBILITY:
Inclusion Criteria:

* opiate dependence
* newly admitted to methadone treatment

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (2):
- United States (2):
  - Institutes for Behavior Resources REACH, Baltimore, Maryland
  - University of Maryland Drug Treatment Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell SG, Monico LB, Lertch E, Kelly SM, Gryczynski J, Jaffe JH, O'Grady KE, Schwartz RP. Counseling Staff's Views of Patient-Centered Methadone Treatment: Changing Program Rules and Staff Roles. J Behav Health Serv Res. 2018 Jul;45(3):506-515. doi: 10.1007/s11414-018-9603-1. PMID 29536342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Started | 149 | 151
Completed | 146 | 149
Not Completed | 3 | 2
Not completed — withdrawn from study | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual | Total
Number analyzed (Participants) | 146 | 149 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.3) | 42.0 (9.8) | 42.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 67 | 121
  Male | 92 | 82 | 174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 90 | 81 | 171
  White | 56 | 66 | 122
  Hispanic | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 146 | 149 | 295

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Opiate Positive Urine Tests
Description: Number of participants with opiate positive urine tests
Time Frame: 12-months post-baseline
Population: Missing data were counted as positive
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
Participants | 89 | 90
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.92, Mixed Models Analysis

2. Secondary Outcome: Number of Participants With Cocaine Positive Urine Tests
Description: Cocaine positive urine drug test
Time Frame: 12-months post-baseline
Population: Missing data were considered positive
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
Participants | 67 | 85
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.06, Mixed Models Analysis

3. Secondary Outcome: Drug Use HIV Risk Behavior
Description: HIV Drug Use Risk Assessment Battery Score ranges from 0 to 22. A higher score is considered to be associated with higher risk.
Time Frame: 12-months post-baseline
Population: Baseline values were used when 12 month data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
units on a scale | 0.72 (2.56) | 1.36 (3.63)
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.08, Mixed Models Analysis

4. Secondary Outcome: Criminal Behavior
Description: Days of criminal behavior
Time Frame: 12-months post-baseline
Measure: Mean (Standard Deviation); unit: Number of Days in the Past 30 days
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
Number of Days in the Past 30 days | 2.99 (.75) | 3.72 (.93)
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.54, Mixed Models Analysis

5. Secondary Outcome: Global Score on the World Health Organization Quality of Life Measure
Description: Scale from 1 through 5. A higher score reflects a better quality of life.
Time Frame: 12-months post-baseline
Population: Baseline values were used when 12 month data were missing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
units on a scale | 3.70 (0.91) | 3.47 (1.0)
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = .04, Mixed Models Analysis

6. Secondary Outcome: Number of Participants Meeting DSM-IV Opiate Dependence Criteria
Description: Diagnostic and Statistical Manual (DSM)-IV criteria for opiate dependence
Time Frame: 12-months post-baseline
Population: Baseline values were used when 12 month data were missing
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
Participants | 88 | 103
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.11, Mixed Models Analysis

7. Secondary Outcome: Number of Participants Meeting DSM-IV Cocaine Dependence Criteria
Description: Number of participants meeting DSM-IV cocaine dependence criteria
Time Frame: 12-months post-baseline
Population: Baseline values were used when 12 month data were missing
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
Number analyzed (Participants) | 146 | 149
Participants | 41 | 52
Statistical Analysis 1: Comparison: Patient-Centered Methadone Treatment vs Methadone Treatment as Usual; Test type: Superiority; p = 0.21, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 year
Description: All Serious Adverse Events were considered unrelated to study participation.
Arm/Group | Patient-Centered Methadone Treatment | Methadone Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 2/146 | 4/149
Serious Adverse Events (participants affected / at risk) | 31/146 | 36/149
Other Adverse Events (participants affected / at risk) | 0/146 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient-Centered Methadone Treatment (N=146) | Methadone Treatment as Usual (N=149)
Pain in Back, Hip, Jaw, Groin (Musculoskeletal and connective tissue disorders) | 3 | 0
Soft Tissue Infection (Infections and infestations) | 6 | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Knee Surgery (Surgical and medical procedures) | 1 | 0
Seizures (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 2 | 4
Hypertension (Vascular disorders) | 4 | 1
Fibroids (Reproductive system and breast disorders) | 1 | 0
Trauma (Injury, poisoning and procedural complications) | 3 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Pancreatitis (Endocrine disorders) | 1 | 0
Lupus (Immune system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Dehydration (General disorders) | 0 | 1
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 3 | 1
Angina (Cardiac disorders) | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 1 | 0
Stroke (Vascular disorders) | 2 | 1
HIV (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 3
Spontaneous abortion (Reproductive system and breast disorders) | 1 | 1
Pulmonary Embolism (Vascular disorders) | 1 | 2
Diabetes Mellitus (Endocrine disorders) | 1 | 1
Altered Mental Status (Nervous system disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 2
Psychiatric Disorder Unspecified (Psychiatric disorders) | 0 | 3
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Kidney stone (Renal and urinary disorders) | 0 | 1
Kidney Infection (Renal and urinary disorders) | 0 | 1
Varices (Vascular disorders) | 0 | 1
Infected catheter (Injury, poisoning and procedural complications) | 0 | 1
Ulcer (Gastrointestinal disorders) | 0 | 1
Edema (Vascular disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Poisoning of Unknown Origin and Type (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes